CLINICAL TRIAL: NCT04798027
Title: Immunogenicity and Safety of the First-in-Human SARS-CoV-2 mRNA Vaccine Formulation in Healthy Adults 18 Years of Age and Older
Brief Title: Study of mRNA Vaccine Formulation Against COVID-19 in Healthy Adults 18 Years of Age and Older
Acronym: VAW00001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision not to pursue further development of this product given the wide availability of authorized/approved mRNA COVID-19 vaccines
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAW00001; U1111-1251-5486 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This was a sequential group prevention study consisting of a sentinel cohort followed by the Full Enrollment Cohort. There were 3 dose levels (up to 25 participants 18-49 years of age for each dose level) in the Sentinel Cohort, which were done in an open-label fashion with stepwise safety evaluation for each dose level and each vaccination. All sentinel participants received 2 vaccinations, 21 days apart. For the Full Enrollment Cohort (FEC), which was done in a double-blind design participants were stratified into 2 groups based on age at enrollment: the younger adult age group (140 planned participants 18-49 years of age) and the older adult age group (168 planned participants greater than or equal to [>=] 50 years of age). The FEC Cohort 1 (Groups 1 to 3) received a single injection of study intervention while participants in Cohort 2 (Groups 4 to 6) received 2 vaccinations (to be given 21 days apart).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the FEC: blinding for vaccine group assignment (formulation) of participants, outcome assessors, Investigators, laboratory personnel, and Sponsor study staff. Only study site staff who prepare and administer the vaccine and were not involved with the safety evaluations were unblinded to vaccine group assignment. There was no blinding for injection schedule.
  The Sentinel Cohort was open-label (no blinding).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Sentinel Cohort: SARS-CoV-2 Vaccine Ultra Low dose (Experimental): Participants received two intramuscular (IM) injections of severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) Vaccine ultra-low dose on Day 1 and at Day 22, respectively.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 1
- Sentinel Cohort: SARS-CoV-2 Vaccine Low dose (Experimental): Participants received two IM injections of SARS-CoV-2 Vaccine low dose on Day 1 and at Day 22, respectively.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 2
- Sentinel Cohort: SARS-CoV-2 Vaccine Medium dose (Experimental): Participants received two IM injections of SARS-CoV-2 Vaccine medium dose on Day 1 and at Day 22, respectively.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 3
- FEC Cohort 1: SARS-CoV-2 Vaccine Ultra Low dose (Experimental): Participants received a single IM injection of SARS-CoV-2 Vaccine ultra-low dose on Day 1.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 1
- FEC Cohort 1: SARS-CoV-2 Vaccine Low dose (Experimental): Participants received a single IM injection of SARS-CoV-2 Vaccine low dose on Day 1.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 2
- FEC Cohort 1: Placebo (Placebo Comparator): Participants received a single IM injection of placebo matched to SARS-CoV-2 Vaccine on Day 1.
  Interventions: Biological: Placebo (0.9% normal saline)
- FEC Cohort 2: SARS-CoV-2 Vaccine Ultra Low dose (Experimental): Participants received two IM injections of SARS-CoV-2 Vaccine ultra-low dose on Day 1 and at Day 22, respectively.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 1
- FEC Cohort 2: SARS-CoV-2 Vaccine Low dose (Experimental): Participants received two IM injections of SARS-CoV-2 Vaccine low dose on Day 1 and at Day 22, respectively.
  Interventions: Biological: SARS-CoV-2 mRNA vaccine formulation 2
- FEC Cohort 2: Placebo (Placebo Comparator): Participants received two IM injections of placebo matched to SARS-CoV-2 Vaccine on Day 1 and at Day 22, respectively.
  Interventions: Biological: Placebo (0.9% normal saline)

INTERVENTIONS:
Biological: SARS-CoV-2 mRNA vaccine formulation 1 — Pharmaceutical form: Sterile suspension Route of administration: Intramuscular injection
  Arms: FEC Cohort 1: SARS-CoV-2 Vaccine Ultra Low dose; FEC Cohort 2: SARS-CoV-2 Vaccine Ultra Low dose; Sentinel Cohort: SARS-CoV-2 Vaccine Ultra Low dose
Biological: SARS-CoV-2 mRNA vaccine formulation 2 — Pharmaceutical form: Sterile suspension Route of administration: Intramuscular injection
  Arms: FEC Cohort 1: SARS-CoV-2 Vaccine Low dose; FEC Cohort 2: SARS-CoV-2 Vaccine Low dose; Sentinel Cohort: SARS-CoV-2 Vaccine Low dose
Biological: SARS-CoV-2 mRNA vaccine formulation 3 — Pharmaceutical form: Sterile suspension Route of administration: Intramuscular injection
  Arms: Sentinel Cohort: SARS-CoV-2 Vaccine Medium dose
Biological: Placebo (0.9% normal saline) — Pharmaceutical form: Liquid Route of administration: Intramuscular injection
  Arms: FEC Cohort 1: Placebo; FEC Cohort 2: Placebo

SUMMARY:
The primary objectives of the study are:

* To describe the safety profile of all participants in each age group and each study intervention group up to 12 months post-last dose.
* To describe the neutralizing antibody profile at Day 1, Day 22, and Day 36 of each study intervention group.

The secondary objectives of the study are:

* To describe binding antibody profile from Day 1 to Day 387 of each study intervention group.
* To describe the neutralizing antibody profile from Day 91 to Day 387 of each study intervention group.
* To describe the occurrence of virologically-confirmed coronavirus disease-2019 (COVID-19)-like illness and serologically-confirmed SARS-CoV-2 infection.
* To evaluate the correlation/association between antibody responses to SARS-CoV-2 messenger RNA (mRNA) vaccine and the risk of virologically-confirmed COVID-19-like illness and/or serologically-confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection.

DETAILED DESCRIPTION:
The duration of each participant's participation in the study was approximately 365 days post-last injection: approximately 386 days duration for participants receiving 2 injections and approximately 365 days duration total for participants receiving a single injection.

ELIGIBILITY:
Inclusion criteria:

* Aged >= 18 years on the day of inclusion.
* A female participant was eligible to participate if she was not pregnant or breastfeeding and one of the following conditions applies:
* Was of non-childbearing potential. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile.

OR

* Was of childbearing potential and agreed to use an effective contraceptive method or abstinence from at least 4 weeks prior to the first vaccination until at least 12 weeks after the last vaccination.

A participant of childbearing potential must had a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours before the study intervention.

* Informed Consent Form had been signed and dated.
* Participant not eligible to receive, based on local guidance, or if eligible does not intend to receive an authorized/approved COVID-19 vaccine from first vaccination until completion of the key timepoint of Day 43 of follow-up of this study.

Exclusion criteria:

* History of COVID-19 disease or prior SARS-CoV-2 infection confirmed serologically.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Chronic illness or condition considered to potentially increase the risk for severe COVID illness or that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion.
* Known liver disease or fatty liver.
* Positive test for chronic active Hepatitis B surface antigen, Hepatitis B core antibody, Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody from blood work collected at screening visit.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination based on Investigator's judgment.
* Receipt of immunoglobulins, blood or blood-derived products in the past 3 months.
* Prior administration of a coronavirus vaccine (SARS-CoV-2, SARS-CoV, Middle East Respiratory Syndrome coronavirus [MERS-CoV]).
* Receipt of any vaccine in the 30 days preceding the first study vaccination or planned receipt of any vaccine in the 30 days following the last study vaccination except for influenza vaccination, which might be received at least 2 weeks before and a minimum of 2 weeks after study vaccines.
* Receipt of any therapy known to have in-vitro antiviral activity against SARS-CoV-2 within 72 hours prior to the first blood draw or planned use of such therapy 72 hours prior to study immunogenicity blood draws at Day 22 and Day 36.
* Residence in a nursing home or long-term care facility.
* Health care workers providing direct patient care for COVID-19 participants.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- United States (12):
  - Investigational Site Number :8400003, Rolling Hills Estates, California
  - Investigational Site Number :8400002, Hollywood, Florida
  - Investigational Site Number :8400006, Miami, Florida
  - Investigational Site Number :8400017, Iowa City, Iowa
  - Investigational Site Number :8400007, Kansas City, Missouri
  - Investigational Site Number :8400008, Omaha, Nebraska
  - Investigational Site Number :8400001, Rochester, New York
  - Investigational Site Number :8400010, Philadelphia, Pennsylvania
  - Investigational Site Number :8400004, North Charleston, South Carolina
  - Investigational Site Number :8400015, Knoxville, Tennessee
  - Investigational Site Number :8400009, Houston, Texas
  - Investigational Site Number :8400005, Salt Lake City, Utah
- Australia (4):
  - Investigational Site Number :0360003, Morayfield, Queensland
  - Investigational Site Number :0360005, South Brisbane, Queensland
  - Investigational Site Number :0360001, Melbourne, Victoria
  - Investigational Site Number :0360002, Nedlands, Western Australia
- Brazil (3):
  - Investigational Site Number :0760001, Salvador, Estado de Bahia
  - Investigational Site Number :0760004, Campo Grande, Mato Grosso do Sul
  - Investigational Site Number :0760003, Belo Horizonte, Minas Gerais
- Honduras (2):
  - Investigational Site Number :3400002, Barrio del Centro
  - Investigational Site Number :3400001, San Pedro Sula

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAW00001 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25380&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 active sites in 4 countries between 12 Mar 2021 and 27 Jun 2022. Study consisted of 2 cohorts: Sentinel Cohort and Full Enrollment Cohort (FEC). For analysis purpose, Baseline, safety and outcome measure data was planned to be collected, analyzed and reported for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Pre-assignment Details: Participants (aged 18-49 years) in Sentinel Cohort received two vaccinations, 21 days apart. FEC participants were stratified into 2 age groups: younger adult group (18-49 years) and the older adult group (greater than or equal to [>=] 50 years). FEC Cohort 1 participants received a single injection of study vaccine or placebo, while participants in Cohort 2 received two vaccinations (21 days apart). A total of 182 participants were enrolled, of which 180 were vaccinated in the study.
Period: Overall Study
Arm/Group | Sentinel Cohort: SARS-CoV-2 Vaccine Ultra Low Dose | Sentinel Cohort: SARS-CoV-2 Vaccine Low Dose | Sentinel Cohort: SARS-CoV-2 Vaccine Medium Dose | FEC Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | FEC Cohort 1: SARS-CoV-2 Vaccine Low Dose | FEC Cohort 1: Placebo | FEC Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | FEC Cohort 2: SARS-CoV-2 Vaccine Low Dose | FEC Cohort 2: Placebo
Started | 10 | 25 | 10 | 27 | 26 | 13 | 28 | 29 | 14
Vaccinated on Day 1 | 10 | 25 | 10 | 27 | 25 | 13 | 28 | 28 | 14
Vaccinated on Day 22 | 10 | 24 | 10 | 0 (Only FEC Cohort 2 participants received second dose of study vaccine at Day 22.) | 0 (Only FEC Cohort 2 participants received second dose of study vaccine at Day 22.) | 0 (Only FEC Cohort 2 participants received second dose of study vaccine at Day 22.) | 19 | 19 | 9
Safety Analysis Set (SafAS) (Participants who had received at least one injection of study intervention and were analyzed according to the study intervention they actually received.) | 18 (8 participants of 'Sentinel Cohort: SARS-CoV-2 Vaccine low dose' received ultra-low dose and were included in arm 'Sentinel Cohort: SARS-CoV-2 Vaccine ultra-low dose' for safety analysis.) | 17 | 10 | 36 (9 participants of 'FEC Cohort 2: SARS-CoV-2 Vaccine ultra-low dose' received ultra-low dose in arm 'FEC Cohort 1: SARS-CoV-2 Vaccine ultra-low dose' and were included in that arm for safety analysis.) | 34 (9 participants of 'FEC Cohort 2: SARS-CoV-2 Vaccine low dose' received low dose in arm 'FEC Cohort 1: SARS-CoV-2 Vaccine low dose' and were included in that arm for safety analysis.) | 18 (5 participants of 'FEC Cohort 2: Placebo' received dose in FEC Cohort 1: Placebo and were included in that arm for safety analysis.) | 19 | 19 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 25 | 10 | 27 | 26 | 13 | 28 | 29 | 14
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 2 | 2
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Sponsor | 8 | 22 | 9 | 26 | 24 | 11 | 25 | 26 | 11

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants according to the intervention to which they were randomized. Data for baseline characteristics was planned to be collected and analyzed for combined population (Full Enrollment Cohort + Sentinel Cohort) in which the same dose-level groups in Sentinel Cohort and Full Enrollment Cohort were pooled for the analysis. Since Sentinel Cohort: SARS-CoV-2 Vaccine Medium Dose group received 2 injections; they were presented under Cohort 2 for analysis.
Groups:
- Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose: Participants received a single IM injection of SARS-CoV-2 Vaccine ultra-low dose on Day 1.
- Cohort 1: SARS-CoV-2 Vaccine Low Dose: Participants received a single IM injection of SARS-CoV-2 Vaccine low dose on Day 1.
- Cohort 1: Placebo: Participants received a single IM injection of placebo matched to SARS-CoV-2 Vaccine on Day 1.
- Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose: Participants received two IM injections of SARS-CoV-2 Vaccine ultra-low dose on Day 1 and at Day 22, respectively.
- Cohort 2: SARS-CoV-2 Vaccine Low Dose: Participants received two IM injections of SARS-CoV-2 Vaccine low dose on Day 1 and at Day 22, respectively.
- Cohort 2: SARS-CoV-2 Vaccine Medium Dose: Participants received two IM injections of SARS-CoV-2 Vaccine medium dose on Day 1 and at Day 22, respectively.
- Cohort 2: Placebo: Participants received two IM injections of placebo matched to SARS-CoV-2 Vaccine on Day 1 and at Day 22, respectively.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo | Total
Number analyzed (Participants) | 27 | 26 | 13 | 38 | 54 | 10 | 14 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.15 (16.19) | 41.96 (17.05) | 39.77 (14.96) | 36.21 (13.00) | 34.96 (13.22) | 31.00 (8.94) | 38.79 (16.24) | 38.01 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 5 | 18 | 25 | 3 | 6 | 77
  Male | 17 | 16 | 8 | 20 | 29 | 7 | 8 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 3 | 12 | 7 | 10 | 3 | 45
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3
  Black or African American | 0 | 2 | 0 | 2 | 8 | 0 | 4 | 16
  White | 22 | 18 | 10 | 24 | 34 | 0 | 5 | 113
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Immediate Unsolicited Adverse Events (AEs)
Description: AE: any untoward medical occurrence in clinical investigation participant administered medicinal product & which did not have any causal relationship with the treatment. Unsolicited AE: observed AE that did not fulfill conditions prelisted in case report form (CRF) in terms of diagnosis &/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, & any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in CRF. Reported AEs were presented as pre-specified in protocol. In the data table, '0' in number analyzed field denotes that no participants were available for assessment for specified Group as no one in that group received vaccination 2.
Time Frame: Within 30 minutes post any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 22])
Population: SafAS: participants who received at least one injection of study vaccine were analyzed by the intervention they actually received. Data were collected & analyzed for the combined population in which same dose-level groups in Sentinel Cohort and FEC were pooled. One ultra-low dose Sentinel Cohort participant who was supposed to receive 2 doses received only 1 & was counted into Cohort 1: ultra-low dose (N = 37; 1 from sentinel cohort and 36 from FEC cohort 1) based on actual injection scheme.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Group 3: Placebo: Participants received a single IM injection of placebo matched to SARS-CoV-2 Vaccine on Day 1.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Group 3: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 37 | 34 | 18 | 36 | 36 | 10 | 9
Participants
  Post Any vaccination | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Post vaccination 2 |  |  |  | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: Solicited reaction (SR): expected adverse reaction (sign or symptom) observed & reported under conditions (nature & onset) prelisted (i.e., solicited) in CRF and considered as related to product administered. Solicited injection site reactions included pain, erythema, & swelling. Reported AEs for each arm were presented as pre-specified in study protocol. In the data table, '0' in number analyzed field denotes that no participants were available for assessment for specified Group as no one in that group received vaccination 2.
Time Frame: Within 7 days after any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 22])
Population: SafAS population. Here, "overall number of participants analyzed" = participants with available data for this outcome measure (OM). Data were collected & analyzed for the combined population in which same dose-level groups in Sentinel Cohort and FEC were pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 36 | 33 | 18 | 36 | 36 | 10 | 9
Participants
  Pain Post-any vaccination | 28 | 28 | 5 | 33 | 33 | 10 | 2
  Pain Post-vaccination 1 | 28 | 28 | 5 | 29 | 32 | 10 | 1
  Pain Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Pain Post-vaccination 2 |  |  |  | 28 | 32 | 10 | 2
  Erythema Post-any vaccination | 2 | 0 | 0 | 4 | 5 | 0 | 0
  Erythema Post-vaccination 1 | 2 | 0 | 0 | 3 | 5 | 0 | 0
  Erythema Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Erythema Post-vaccination 2 |  |  |  | 2 | 4 | 0 | 0
  Swelling Post-any vaccination | 1 | 2 | 0 | 6 | 4 | 2 | 0
  Swelling Post-vaccination 1 | 1 | 2 | 0 | 3 | 3 | 2 | 0
  Swelling Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Swelling Post-vaccination 2 |  |  |  | 4 | 2 | 1 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: SR was an expected adverse reaction (sign or symptom) observed & reported under conditions (nature & onset) prelisted (i.e., solicited) in CRF & considered as related to product administered. Solicited systemic reactions included fever, headache, malaise, myalgia, arthralgia & chills. Reported AEs for each arm were presented as pre-specified in study protocol. In the data table, '0' in number analyzed field denotes that no participants were available for assessment for specified Group as no one in that group received vaccination 2.
Time Frame: Within 7 days after any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 22])
Population: SafAS population. Here, "overall number of participants analyzed" = participants with available data for this OM. Data were collected & analyzed for the combined population in which same dose-level groups in Sentinel Cohort and FEC were pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 36 | 33 | 18 | 36 | 36 | 10 | 9
Participants
  Fever Post-any vaccination: number analyzed (Participants) | 35 | 33 | 18 | 36 | 36 | 10 | 9
  Fever Post-any vaccination | 5 | 8 | 1 | 9 | 16 | 10 | 0
  Fever Post-vaccination 1: number analyzed (Participants) | 35 | 33 | 18 | 36 | 36 | 10 | 9
  Fever Post-vaccination 1 | 5 | 8 | 1 | 6 | 11 | 10 | 0
  Fever Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 34 | 36 | 10 | 9
  Fever Post-vaccination 2 |  |  |  | 7 | 12 | 8 | 0
  Headache Post-any vaccination | 17 | 17 | 6 | 26 | 31 | 10 | 5
  Headache Post-vaccination 1 | 17 | 17 | 6 | 22 | 27 | 9 | 3
  Headache Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Headache Post-vaccination 2 |  |  |  | 21 | 27 | 7 | 3
  Malaise Post-any vaccination | 21 | 21 | 5 | 28 | 31 | 10 | 2
  Malaise Post-vaccination 1 | 21 | 21 | 5 | 25 | 28 | 9 | 2
  Malaise Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Malaise Post-vaccination 2 |  |  |  | 22 | 28 | 9 | 2
  Myalgia Post-any vaccination | 20 | 23 | 4 | 28 | 28 | 8 | 2
  Myalgia Post-vaccination 1 | 20 | 23 | 4 | 23 | 24 | 8 | 2
  Myalgia Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Myalgia Post-vaccination 2 |  |  |  | 22 | 25 | 7 | 2
  Arthralgia Post-any vaccination | 7 | 13 | 2 | 20 | 23 | 10 | 2
  Arthralgia Post-vaccination 1 | 7 | 13 | 2 | 11 | 18 | 5 | 1
  Arthralgia Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Arthralgia Post-vaccination 2 |  |  |  | 17 | 19 | 7 | 2
  Chills Post-any vaccination | 14 | 17 | 4 | 20 | 29 | 9 | 1
  Chills Post-vaccination 1 | 14 | 17 | 4 | 15 | 23 | 8 | 0
  Chills Post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Chills Post-vaccination 2 |  |  |  | 17 | 25 | 7 | 1

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which did not have any casual relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination. Reported AEs for each arm were presented as pre-specified in the study protocol. In the data table, '0' in number analyzed field denotes that no participants were available for assessment for specified Group as no one in that group received vaccination 2.
Time Frame: Within 21 days after any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 22])
Population: Analyzed on SafAS population. Data were collected & analyzed for the combined population in which same dose-level groups in Sentinel Cohort and FEC were pooled. One ultra-low dose Sentinel Cohort participant who was supposed to receive 2 doses received only 1 & was counted into Cohort 1: ultra-low dose (N = 37; 1 from sentinel cohort and 36 from FEC cohort 1) based on actual injection scheme.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 37 | 34 | 18 | 36 | 36 | 10 | 9
Participants
  Post Any vaccination | 17 | 4 | 8 | 10 | 15 | 5 | 3
  Post vaccination 1 | 17 | 4 | 8 | 10 | 10 | 5 | 2
  Post vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 36 | 36 | 10 | 9
  Post vaccination 2 |  |  |  | 5 | 10 | 2 | 1

5. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs), Adverse Event of Special Interest (AESIs) and Medically Attended Adverse Events (MAAEs)
Description: SAEs: any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. AESIs: event for which ongoing monitoring & rapid communication by investigator to the sponsor was done. MAAE was a new onset or worsening of a condition that prompted participant or participant's parent/legally acceptable representative to seek unplanned medical advice at physician's office or emergency department. Reported AEs for each arm were presented as pre-specified in study protocol.
Time Frame: From Day 1 until 12 months post last vaccination (i.e., up to Day 366 for Cohort 1 groups and up to Day 387 for Cohort 2 groups)
Population: Analysis was performed on SafAS population. Data were collected & analyzed for the combined population in which same dose-level groups in Sentinel Cohort and FEC were pooled. One ultra-low dose Sentinel Cohort participant who was supposed to receive 2 doses received only 1 & was counted into Cohort 1: ultra-low dose (N = 37; 1 from sentinel cohort and 36 from FEC cohort 1) based on actual injection scheme.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 37 | 34 | 18 | 36 | 36 | 10 | 9
Participants
  SAEs | 0 | 0 | 1 | 0 | 0 | 1 | 0
  AESI | 3 | 3 | 2 | 3 | 1 | 1 | 1
  MAAEs | 6 | 2 | 1 | 6 | 6 | 3 | 2

6. Primary Outcome: Number of Participants With Laboratory Test Results Based on US Food and Drug Administration (FDA) Toxicity Grading Guidance
Description: Laboratory tests: hemoglobin (male & female), above & below normal white blood cell, lymphocytes, neutrophils & eosinophils, platelet count, creatinine & blood urea nitrogen, hyponatremia & hypernatremia, hyperkalemia & hypokalemia, hyperglycemia (non-fasting), hypoproteinemia, alkaline phosphate, alanine aminotransferase, aspartate aminotransferase, bilirubin (with any increase in liver function test [LFT], bilirubin (normal LFT), prothrombin & partial thromboplastin time (seconds), Urine: protein, glucose & blood. US FDA "Toxicity Grading Scale for Healthy Adults & Adolescent Volunteers" was used for grading; Grade 1=mild, Grade 2=moderate & Grade 3=severe. In the data table, 'number analyzed'=participants with available data for each specified category & '0'=none of participants were available for assessment for specified Group.
Time Frame: From Day 1 up to up to 8 days post last vaccination (i.e., up to Day 9 for Cohort 1 groups; up to Day 30 for Cohort 2 groups)
Population: SafAS. "Overall number of participants analyzed" = participants with available data for this OM. Data were collected & analyzed for the combined population in which same dose-level groups in Sentinel Cohort and FEC were pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 35 | 33 | 18 | 33 | 36 | 10 | 9
Participants
  Hemoglobin (Female): Grade 1: number analyzed (Participants) | 13 | 14 | 6 | 16 | 15 | 3 | 5
  Hemoglobin (Female): Grade 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1
  Hemoglobin (Female): Grade 2: number analyzed (Participants) | 13 | 14 | 6 | 16 | 15 | 3 | 5
  Hemoglobin (Female): Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hemoglobin (Female): Grade 3: number analyzed (Participants) | 13 | 14 | 6 | 16 | 15 | 3 | 5
  Hemoglobin (Female): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (Male): Grade 1: number analyzed (Participants) | 22 | 19 | 12 | 17 | 20 | 7 | 4
  Hemoglobin (Male): Grade 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
  Hemoglobin (Male): Grade 2: number analyzed (Participants) | 22 | 19 | 12 | 17 | 20 | 7 | 4
  Hemoglobin (Male): Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (Male): Grade 3: number analyzed (Participants) | 22 | 19 | 12 | 17 | 20 | 7 | 4
  Hemoglobin (Male): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Above normal white blood cell: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Above normal white blood cell: Grade 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Above normal white blood cell: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Above normal white blood cell: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Above normal white blood cell: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Above normal white blood cell: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Below normal white blood cell: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Below normal white blood cell: Grade 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1
  Below normal white blood cell: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Below normal white blood cell: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Below normal white blood cell: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Below normal white blood cell: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decreased: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Platelets Decreased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decreased: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Platelets Decreased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decreased: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Platelets Decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Neutrophils Decreased: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Neutrophils Decreased: Grade 1 | 1 | 1 | 1 | 0 | 6 | 0 | 0
  Absolute Neutrophils Decreased: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Neutrophils Decreased: Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Absolute Neutrophils Decreased: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Neutrophils Decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Lymphocytes Decreased: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Lymphocytes Decreased: Grade 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Absolute Lymphocytes Decreased: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Lymphocytes Decreased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Lymphocytes Decreased: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Lymphocytes Decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Eosinophils: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Eosinophils: Grade 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Absolute Eosinophils: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Eosinophils: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Eosinophils: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 33 | 35 | 10 | 9
  Absolute Eosinophils: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 1: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hyponatremia: Grade 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0
  Hyponatremia: Grade 2: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hyponatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hyponatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hypernatremia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hypernatremia: Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hypernatremia: Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hyperkalemia: Grade 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Hyperkalemia: Grade 2: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hyperkalemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 3: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hyperkalemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hypokalemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hypokalemia: Grade 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Hypokalemia: Grade 3: number analyzed (Participants) | 35 | 32 | 18 | 32 | 35 | 10 | 9
  Hypokalemia: Grade 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Blood Urea Nitrogen: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Blood Urea Nitrogen: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Blood Urea Nitrogen: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Creatinine: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Creatinine: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Creatinine: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Hyperglycemia: Grade 1 | 2 | 0 | 0 | 2 | 3 | 0 | 0
  Hyperglycemia: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Hyperglycemia: Grade 2 | 2 | 0 | 0 | 1 | 2 | 0 | 0
  Hyperglycemia: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Hyperglycemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoproteinemia: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Hypoproteinemia: Grade 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Hypoproteinemia: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Hypoproteinemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoproteinemia: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Hypoproteinemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Alanine aminotransferase: Grade 1 | 1 | 0 | 2 | 0 | 1 | 2 | 0
  Alanine aminotransferase: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Alanine aminotransferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Alanine aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Aspartate aminotransferase: Grade 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0
  Aspartate aminotransferase: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Aspartate aminotransferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Aspartate aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphate: Grade 1: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Alkaline phosphate: Grade 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  Alkaline phosphate: Grade 2: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Alkaline phosphate: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphate: Grade 3: number analyzed (Participants) | 35 | 33 | 18 | 32 | 35 | 10 | 9
  Alkaline phosphate: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin - with any increase in LFT: Grade 1: number analyzed (Participants) | 2 | 0 | 3 | 0 | 1 | 2 | 0
  Bilirubin - with any increase in LFT: Grade 1 | 0 |  | 0 |  | 0 | 0 |
  Bilirubin - with any increase in LFT: Grade 2: number analyzed (Participants) | 2 | 0 | 3 | 0 | 1 | 2 | 0
  Bilirubin - with any increase in LFT: Grade 2 | 0 |  | 0 |  | 0 | 0 |
  Bilirubin - with any increase in LFT: Grade 3: number analyzed (Participants) | 2 | 0 | 3 | 0 | 1 | 2 | 0
  Bilirubin - with any increase in LFT: Grade 3 | 0 |  | 0 |  | 0 | 0 |
  Bilirubin - with normal in LFT: Grade 1: number analyzed (Participants) | 33 | 33 | 15 | 32 | 34 | 8 | 9
  Bilirubin - with normal in LFT: Grade 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin - with normal in LFT: Grade 2: number analyzed (Participants) | 33 | 33 | 15 | 32 | 34 | 8 | 9
  Bilirubin - with normal in LFT: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin - with normal in LFT: Grade 3: number analyzed (Participants) | 33 | 33 | 15 | 32 | 34 | 8 | 9
  Bilirubin - with normal in LFT: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin time: Grade 1: number analyzed (Participants) | 33 | 32 | 18 | 32 | 34 | 10 | 9
  Prothrombin time: Grade 1 | 0 | 2 | 0 | 3 | 3 | 0 | 0
  Prothrombin time: Grade 2: number analyzed (Participants) | 33 | 32 | 18 | 32 | 34 | 10 | 9
  Prothrombin time: Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Prothrombin time: Grade 3: number analyzed (Participants) | 33 | 32 | 18 | 32 | 34 | 10 | 9
  Prothrombin time: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial thromboplastin time: Grade 1: number analyzed (Participants) | 32 | 30 | 17 | 32 | 34 | 10 | 9
  Partial thromboplastin time: Grade 1 | 1 | 2 | 1 | 3 | 2 | 0 | 0
  Partial thromboplastin time: Grade 2: number analyzed (Participants) | 32 | 30 | 17 | 32 | 34 | 10 | 9
  Partial thromboplastin time: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial thromboplastin time: Grade 3: number analyzed (Participants) | 32 | 30 | 17 | 32 | 34 | 10 | 9
  Partial thromboplastin time: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine - glucose: Grade 1: number analyzed (Participants) | 33 | 33 | 17 | 32 | 36 | 10 | 8
  Urine - glucose: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine - glucose: Grade 2: number analyzed (Participants) | 33 | 33 | 17 | 32 | 36 | 10 | 8
  Urine - glucose: Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine - glucose: Grade 3: number analyzed (Participants) | 33 | 33 | 17 | 32 | 36 | 10 | 8
  Urine - glucose: Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine - protein: Grade 1: number analyzed (Participants) | 33 | 33 | 17 | 32 | 36 | 10 | 8
  Urine - protein: Grade 1 | 3 | 5 | 2 | 1 | 4 | 1 | 1
  Urine - protein: Grade 2: number analyzed (Participants) | 33 | 33 | 17 | 32 | 36 | 10 | 8
  Urine - protein: Grade 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Urine - protein: Grade 3: number analyzed (Participants) | 33 | 33 | 17 | 32 | 36 | 10 | 8
  Urine - protein: Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine - blood: Grade 1: number analyzed (Participants) | 7 | 4 | 3 | 11 | 5 | 3 | 3
  Urine - blood: Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Urine - blood: Grade 2: number analyzed (Participants) | 7 | 4 | 3 | 11 | 5 | 3 | 3
  Urine - blood: Grade 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Urine - blood: Grade 3: number analyzed (Participants) | 7 | 4 | 3 | 11 | 5 | 3 | 3
  Urine - blood: Grade 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0

7. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine at Day 1
Description: GMTs of SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Titers were expressed in terms of 1/dilution. Data for this OM was planned to be collected and analyzed for combined population (FEC+ Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: Day 1 (pre-vaccination)
Population: Analyzed on modified full analysis set (mFAS) population that included all participants who received at least one injection of study intervention, analyzed according to the intervention they actually received, and excludes participants with positive pseudovirus neutralization test results against SARS-CoV-2 D614G variant at Baseline (Day 1). Here, "overall number of participants analyzed" signifies participants with available data for this OM.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 34 | 28 | 16 | 32 | 32 | 10 | 8
titer | 5.00 [NA to NA] — 95% confidence interval (CI) was not computable as the standard deviation (SD) of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

8. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine at Day 22
Description: GMTs of SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Titers were expressed in terms of 1/dilution.
Time Frame: Day 22 (post-vaccination)
Population: Analyzed on mFAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM. Data for this OM was planned to be collected and analyzed for combined population (FEC+ Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 31 | 24 | 16 | 32 | 31 | 10 | 9
titer | 24.0 [15.3 to 37.6] | 29.7 [14.8 to 59.6] | 6.66 [3.61 to 12.3] | 35.2 [21.0 to 59.0] | 27.7 [16.4 to 46.9] | 68.2 [29.0 to 160] | 12.8 [2.52 to 65.1]

9. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine at Day 36
Description: as for outcome 8
Time Frame: Day 36 (post-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Cohort 1: Group 2: SARS-CoV-2 Vaccine Low Dose: Participants received a single IM injection of SARS-CoV-2 Vaccine low dose on Day 1.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: Group 2: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 25 | 18 | 13 | 29 | 31 | 10 | 9
titer | 13.6 [8.88 to 20.9] | 30.1 [15.5 to 58.6] | 6.48 [3.68 to 11.4] | 174 [111 to 273] | 223 [147 to 336] | 416 [303 to 570] | 11.6 [2.43 to 55.5]

10. Primary Outcome: Geometric Mean Fold-rise (GMFR) of Serum Neutralization Antibody Titers at Day 22
Description: SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Fold-rise was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (Day 22) and pre-vaccination (on Day 1) i.e., Day 22/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 22 (post-vaccination)
Population: Analyzed on mFAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 31 | 24 | 15 | 32 | 31 | 10 | 8
ratio | 4.80 [3.07 to 7.52] | 5.93 [2.95 to 11.9] | 1.36 [0.704 to 2.62] | 7.05 [4.21 to 11.8] | 5.55 [3.28 to 9.37] | 13.6 [5.79 to 32.1] | 1.32 [0.682 to 2.57]

11. Primary Outcome: Geometric Mean Fold-rise of Serum Neutralization Antibody Titers at Day 36
Description: SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Fold-rise was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (Day 36) and pre-vaccination (on Day 1) i.e., Day 36/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 36 (post-vaccination)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- Cohort 1: SARS-CoV-2 Vaccine Low Dose: Participants received a single IM injection of SARS-CoV-2 Vaccine medium dose on Day 1.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 24 | 18 | 12 | 29 | 31 | 10 | 8
ratio | 2.84 [1.83 to 4.40] | 6.03 [3.10 to 11.7] | 1.32 [0.714 to 2.46] | 34.9 [22.3 to 54.6] | 44.6 [29.5 to 67.3] | 83.1 [60.7 to 114] | 1.20 [0.777 to 1.86]

12. Primary Outcome: Percentage of Participants With >=2-fold and >=4-fold Rise in Serum Neutralization Antibody Titers at Day 22
Description: SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. The fold rise (2-fold and 4-fold) was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (on Day 22) and pre-vaccination (on Day 1) i.e., Day 22/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 22 (post-vaccination)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 31 | 24 | 15 | 32 | 31 | 10 | 8
percentage of participants
  >=2-fold rise | 77.4 [58.9 to 90.4] | 66.7 [44.7 to 84.4] | 6.7 [0.2 to 31.9] | 81.3 [63.6 to 92.8] | 74.2 [55.4 to 88.1] | 100 [69.2 to 100] | 12.5 [0.3 to 52.7]
  >=4-fold rise | 58.1 [39.1 to 75.5] | 58.3 [36.6 to 77.9] | 6.7 [0.2 to 31.9] | 71.9 [53.3 to 86.3] | 54.8 [36.0 to 72.7] | 100 [69.2 to 100] | 12.5 [0.3 to 52.7]

13. Primary Outcome: Percentage of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titer at Day 36
Description: SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. The fold rise (2-fold and 4-fold) was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (on Day 36) and pre-vaccination (on Day 1) i.e., Day 36/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 36 (post-vaccination)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: Group 1: SARS-CoV-2 Vaccine Ultra Low Dose: Participants received a single IM injection of SARS-CoV-2 Vaccine ultra-low dose on Day 1.
- Cohort 2: Group 4: SARS-CoV-2 Vaccine Ultra Low Dose: Participants received two IM injections of SARS-CoV-2 Vaccine ultra-low dose on Day 1 and at Day 22, respectively.
- Cohort 2: Group 5: SARS-CoV-2 Vaccine Low Dose: Participants received two IM injections of SARS-CoV-2 Vaccine low dose on Day 1 and at Day 22, respectively.
- Cohort 2: Group 6: SARS-CoV-2 Vaccine Medium Dose: Participants received two IM injections of SARS-CoV-2 Vaccine medium dose on Day 1 and at Day 22, respectively.
- Cohort 2: Group 7: Placebo: Participants received two IM injections of placebo matched to SARS-CoV-2 Vaccine on Day 1 and at Day 22, respectively.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: Group 2: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Group 3: Placebo | Cohort 2: Group 4: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: Group 5: SARS-CoV-2 Vaccine Low Dose | Cohort 2: Group 6: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Group 7: Placebo
Number analyzed (Participants) | 24 | 18 | 12 | 29 | 31 | 10 | 8
percentage of participants
  >=2-fold rise | 58.3 [36.6 to 77.9] | 77.8 [52.4 to 93.6] | 8.3 [0.2 to 38.5] | 96.6 [82.2 to 99.9] | 100 [88.8 to 100] | 100 [69.2 to 100] | 12.5 [0.3 to 52.7]
  >=4-fold rise | 45.8 [25.6 to 67.2] | 66.7 [41.0 to 86.7] | 8.3 [0.2 to 38.5] | 96.6 [82.2 to 99.9] | 100 [88.8 to 100] | 100 [69.2 to 100] | 12.5 [0.3 to 52.7]

14. Primary Outcome: Percentage of Participants Achieving Seroconversion Against SARS-CoV-2 Virus Antigens at Day 22
Description: Seroconversion was defined as participants with a Baseline (Day 1) titer values below lower limit of quantification (LLOQ) with a detectable neutralization antibody titer above assay LLOQ post injection (at Day 22). LLOQ of the neutralization assay was a titer of 10.
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 31 | 24 | 15 | 32 | 31 | 10 | 8
percentage of participants | 77.4 [58.9 to 90.4] | 66.7 [44.7 to 84.4] | 6.7 [0.2 to 31.9] | 81.3 [63.6 to 92.8] | 74.2 [55.4 to 88.1] | 100 [69.2 to 100] | 12.5 [0.3 to 52.7]

15. Primary Outcome: Percentage of Participants Achieving Seroconversion Against SARS-CoV-2 Virus Antigens at Day 36
Description: Seroconversion was defined as participants with a Baseline (Day 1) titer values below LLOQ with a detectable neutralization antibody titer above assay LLOQ post injection (at Day 36). LLOQ of the neutralization assay was a titer of 10.
Time Frame: Day 36 (post-vaccination)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 24 | 18 | 12 | 29 | 31 | 10 | 8
percentage of participants | 58.3 [36.6 to 77.9] | 77.8 [52.4 to 93.6] | 8.3 [0.2 to 38.5] | 96.6 [82.2 to 99.9] | 100 [88.8 to 100] | 100 [69.2 to 100] | 12.5 [0.3 to 52.7]

16. Secondary Outcome: Geometric Mean Concentration (GMC) of Anti-S Binding Antibody at Day 1, 22, 36, 91, 112, 181, and 202
Description: GMC of Anti-S binding antibodies were assessed using enzyme-linked immunosorbent assay (ELISA) and were measured in ELISA unit/mL (ELU/mL). Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: Day 1 (pre-vaccination); Day 22 (post-vaccination), Day 36 (post-vaccination), Day 91 (only for Cohort 1), Day 112 (only for Cohort 2), Day 181 (only for Cohort 1), and Day 202 (only for Cohort 2)
Population: Analyzed on mFAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM and 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were evaluable for assessment in specified Groups for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 34 | 26 | 16 | 32 | 32 | 10 | 9
ELU/mL
  Day 1 | 10.8 [9.08 to 12.7] | 10.8 [8.84 to 13.1] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 10.1 [8.78 to 11.7] | 10.5 [8.93 to 12.3] | 10.3 [8.52 to 12.4] | 14.4 [7.08 to 29.4]
  Day 22: number analyzed (Participants) | 31 | 24 | 16 | 32 | 32 | 10 | 9
  Day 22 | 239 [153 to 375] | 372 [192 to 723] | 13.2 [7.84 to 22.4] | 448 [249 to 805] | 476 [279 to 812] | 1618 [984 to 2660] | 34.5 [5.22 to 228]
  Day 36: number analyzed (Participants) | 25 | 20 | 13 | 29 | 31 | 10 | 9
  Day 36 | 188 [110 to 319] | 310 [165 to 582] | 14.1 [7.52 to 26.3] | 3618 [2431 to 5382] | 4903 [3326 to 7228] | 10952 [7252 to 16540] | 34.4 [5.31 to 223]
  Day 91: number analyzed (Participants) | 8 | 8 | 5 | 0 | 0 | 0 | 0
  Day 91 | 185 [36.4 to 936] | 1122 [117 to 10789] | 31.2 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. |  |  |  |
  Day 112: number analyzed (Participants) | 0 | 0 | 0 | 15 | 23 | 10 | 6
  Day 112 |  |  |  | 4548 [1090 to 18981] | 1435 [696 to 2962] | 2782 [1138 to 6799] | 96.3 [6.61 to 1402]
  Day 181: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181 | 62.8 | 23251 |  |  |  |  |
  Day 202: number analyzed (Participants) | 0 | 0 | 0 | 1 | 14 | 0 | 1
  Day 202 |  |  |  | 384 | 1209 [344 to 4257] |  | 17316

17. Secondary Outcome: Geometric Mean Fold-rise (GMFR) of Binding Antibody Concentration at Day 22, 36, 91, 112, 181, and 202
Description: Binding antibody titers were evaluated by ELISA. Fold-rise was calculated as the ratio of geometric mean concentrations of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., Day 22/Day 1, Day 36/Day 1, Day 91/Day 1, Day 112/Day 1, Day 181/Day 1, and Day 202/Day 1. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: as for outcome 16
Population: Analyzed on mFAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM and, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were evaluable for assessment in the specified Groups for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 31 | 22 | 15 | 32 | 32 | 10 | 9
ratio
  Day 22/Day 1 | 22.5 [13.9 to 36.2] | 36.7 [17.5 to 76.9] | 1.28 [0.757 to 2.15] | 44.2 [24.4 to 80.0] | 45.3 [26.6 to 77.3] | 158 [93.7 to 265] | 2.39 [0.626 to 9.13]
  Day 36/Day 1: number analyzed (Participants) | 24 | 18 | 12 | 29 | 31 | 10 | 9
  Day 36/Day 1 | 19.5 [11.1 to 34.1] | 30.2 [14.6 to 62.7] | 1.34 [0.706 to 2.53] | 354 [228 to 551] | 466 [318 to 682] | 1067 [712 to 1601] | 2.38 [0.645 to 8.81]
  Day 91/Day 1: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91/Day 1 | 26.8 [4.80 to 150] | 135 [9.27 to 1971] | 2.83 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. |  |  |  |
  Day 112/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 23 | 10 | 6
  Day 112/Day 1 |  |  |  | 481 [115 to 2009] | 131 [61.0 to 282] | 271 [110 to 670] | 5.40 [0.445 to 65.5]
  Day 181/Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1 | 6.65 | 2460 |  |  |  |  |
  Day 202/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 14 | 0 | 1
  Day 202/Day 1 |  |  |  | 40.6 | 101 [25.9 to 392] |  | 125

18. Secondary Outcome: Percentage of Participants With >=2- and >=4- Fold Rise in Anti-S Binding Antibody Concentration at Day 22, 36, 91, 112, 181, and 202
Description: Binding antibody titers were evaluated by ELISA. Fold-rise (2-fold and 4-fold) was calculated as the ratio of geometric mean concentrations of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., Day 22/Day 1, Day 36/Day 1, Day 91/Day 1, Day 112/Day 1, Day 181/Day 1, and Day 202/Day 1. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: as for outcome 16
Population: Analyzed on mFAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM, and 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were evaluable for assessment in the specified Groups for the specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 31 | 22 | 15 | 32 | 32 | 10 | 9
percentage of participants
  Day 22/Day 1: >=2-fold rise | 100 [88.8 to 100] | 100 [84.6 to 100] | 6.7 [0.2 to 31.9] | 93.8 [79.2 to 99.2] | 96.9 [83.8 to 99.9] | 100 [69.2 to 100] | 22.2 [2.8 to 60.0]
  Day 22/Day 1: >=4-fold rise | 90.3 [74.2 to 98.0] | 86.4 [65.1 to 97.1] | 6.7 [0.2 to 31.9] | 90.6 [75.0 to 98.0] | 93.8 [79.2 to 99.2] | 100 [69.2 to 100] | 22.2 [2.8 to 60.0]
  Day 36/Day 1: >=2-fold rise: number analyzed (Participants) | 24 | 18 | 12 | 29 | 31 | 10 | 9
  Day 36/Day 1: >=2-fold rise | 95.8 [78.9 to 99.9] | 100 [81.5 to 100] | 8.3 [0.2 to 38.5] | 100 [88.1 to 100] | 100 [88.8 to 100] | 100 [69.2 to 100] | 22.2 [2.8 to 60.0]
  Day 36/Day 1: >=4-fold rise: number analyzed (Participants) | 24 | 18 | 12 | 29 | 31 | 10 | 9
  Day 36/Day 1: >=4-fold rise | 87.5 [67.6 to 97.3] | 88.9 [65.3 to 98.6] | 8.3 [0.2 to 38.5] | 100 [88.1 to 100] | 100 [88.8 to 100] | 100 [69.2 to 100] | 22.2 [2.8 to 60.0]
  Day 91/Day 1: >=2-fold rise: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91/Day 1: >=2-fold rise | 85.7 [42.1 to 99.6] | 100 [59.0 to 100] | 25.0 [0.6 to 80.6] |  |  |  |
  Day 91/Day 1: >=4-fold rise: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91/Day 1: >=4-fold rise | 85.7 [42.1 to 99.6] | 100 [59.0 to 100] | 25.0 [0.6 to 80.6] |  |  |  |
  Day 112/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 15 | 23 | 10 | 6
  Day 112/Day 1: >=2-fold rise |  |  |  | 100 [78.2 to 100] | 100 [85.2 to 100] | 100 [69.2 to 100] | 50.0 [11.8 to 88.2]
  Day 112/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 15 | 23 | 10 | 6
  Day 112/Day 1: >=4-fold rise |  |  |  | 100 [78.2 to 100] | 100 [85.2 to 100] | 100 [69.2 to 100] | 50.0 [11.8 to 88.2]
  Day 181/Day 1: >=2-fold rise: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=2-fold rise | 100 [2.5 to 100] | 100 [2.5 to 100] |  |  |  |  |
  Day 181/Day 1: >=4-fold rise: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=4-fold rise | 100 [2.5 to 100] | 100 [2.5 to 100] |  |  |  |  |
  Day 202/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 1 | 14 | 0 | 1
  Day 202/Day 1: >=2-fold rise |  |  |  | 100 [2.5 to 100] | 100 [76.8 to 100] |  | 100 [2.5 to 100]
  Day 202/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 1 | 14 | 0 | 1
  Day 202/Day 1: >=4-fold rise |  |  |  | 100 [2.5 to 100] | 100 [76.8 to 100] |  | 100 [2.5 to 100]

19. Secondary Outcome: Geometric Mean Titers of Neutralizing Antibody Titer Against SARS-CoV-2 Recombinant Protein Vaccine Formulations at Day 91, 112, 181, and 202
Description: GMTs of SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Titers were expressed in terms of 1/dilution. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: Cohort 1: Day 91, Day 181 and Cohort 2: Day 112, and Day 202 (post-vaccination)
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 8 | 7 | 5 | 15 | 22 | 10 | 6
titers
  Day 91: number analyzed (Participants) | 8 | 7 | 5 | 0 | 0 | 0 | 0
  Day 91 | 13.7 [6.70 to 28.1] | 113 [10.2 to 1263] | 9.33 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. |  |  |  |
  Day 112: number analyzed (Participants) | 0 | 0 | 0 | 15 | 22 | 10 | 6
  Day 112 |  |  |  | 322 [56.3 to 1842] | 69.5 [31.4 to 154] | 177 [52.7 to 593] | 23.1 [2.91 to 183]
  Day 181: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181 | 21.0 | 2993 |  |  |  |  |
  Day 202: number analyzed (Participants) | 0 | 0 | 0 | 1 | 12 | 0 | 1
  Day 202 |  |  |  | 45.0 | 120 [25.5 to 568] |  | 3490

20. Secondary Outcome: Geometric Mean Fold-rise of Serum Neutralization Antibody Titer at Day 91, 112, 181, and 202
Description: SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Fold-rise was calculated as the ratio of titer values of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., for Cohort 1: Day 91/Day 1, Day 181/Day 1; Cohort 2: Day 112/Day 1, and Day 202/Day 1. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: Day 1 (pre-vaccination), Cohort 1: Day 91, Day 181 and Cohort 2: Day 112, and Day 202 (post-vaccination)
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose: Participants received a single IM injection of SARS-CoV-2 Vaccine ultra- low dose on Day 1.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 7 | 4 | 15 | 22 | 10 | 5
ratio
  Day 91/Day 1: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91/Day 1 | 3.17 [1.49 to 6.74] | 22.7 [2.03 to 253] | 2.18 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. |  |  |  |
  Day 112/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 15 | 22 | 10 | 5
  Day 112/Day 1 |  |  |  | 64.4 [11.3 to 368] | 13.9 [6.28 to 30.7] | 35.3 [10.5 to 119] | 2.76 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Day 181/Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1 | 4.20 | 599 |  |  |  |  |
  Day 202/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 12 | 0 | 0
  Day 202/Day 1 |  |  |  | 9.00 | 24.1 [5.09 to 114] |  |

21. Secondary Outcome: Percentage of Participants With 2-Fold and 4-Fold Rise in Serum Neutralization Antibody Titer at Day 91, 112, 181, and 202
Description: SARS-CoV-2 neutralizing antibodies (D614G variant) was measured using a neutralization assay. Fold-rise (2-fold and 4-fold) was calculated as the ratio of geometric mean concentrations of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., Day 91/Day 1, Day 112/Day 1, Day 181/Day 1, and Day 202/Day 1. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: Day 1 (pre-vaccination), Cohort 1: Day 91, Day 181 and Cohort 2: Day 112, and Day 202 (post-vaccination)
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Group 3: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 7 | 4 | 15 | 22 | 10 | 5
percentage of participants
  Day 91/Day 1: >=2-fold rise: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91/Day 1: >=2-fold rise | 71.4 [29.0 to 96.3] | 71.4 [29.0 to 96.3] | 25.0 [0.6 to 80.6] |  |  |  |
  Day 91/Day 1: >=4-fold rise: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91/Day 1: >=4-fold rise | 57.1 [18.4 to 90.1] | 71.4 [29.0 to 96.3] | 25.0 [0.6 to 80.6] |  |  |  |
  Day 112/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 15 | 22 | 10 | 5
  Day 112/Day 1: >=2-fold rise |  |  |  | 93.3 [68.1 to 99.8] | 90.9 [70.8 to 98.9] | 100 [69.2 to 100] | 40.0 [5.3 to 85.3]
  Day 112/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 15 | 22 | 10 | 5
  Day 112/Day 1: >=4-fold rise |  |  |  | 86.7 [59.5 to 98.3] | 77.3 [54.6 to 92.2] | 100 [69.2 to 100] | 20.0 [0.5 to 71.6]
  Day 181/Day 1: >=2-fold rise: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=2-fold rise | 100 [2.5 to 100] | 100 [2.5 to 100] |  |  |  |  |
  Day 181/Day 1: >=4-fold rise: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=4-fold rise | 100 [2.5 to 100] | 100 [2.5 to 100] |  |  |  |  |
  Day 202/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 1 | 12 | 0 | 0
  Day 202/Day 1: >=2-fold rise |  |  |  | 100 [2.5 to 100] | 91.7 [61.5 to 99.8] |  |
  Day 202/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 1 | 12 | 0 | 0
  Day 202/Day 1: >=4-fold rise |  |  |  | 100 [2.5 to 100] | 83.3 [51.6 to 97.9] |  |

22. Secondary Outcome: Percentage of Participants Achieving Seroconversion Against SARS-CoV-2 Virus Antigens
Description: Seroconversion was defined as participants with a Baseline (Day 1) titer values below lower limit of quantification (LLOQ) with a detectable neutralization antibody titer above assay LLOQ post injection. LLOQ of the neutralization assay was a titer of 10. Data for this OM was planned to be collected and analyzed for combined population (FEC + Sentinel Cohort) in which same dose-level groups in Sentinel Cohort and FEC were pooled for analysis.
Time Frame: Cohort 1: Day 91, Day 181 and Cohort 2: Day 112, and Day 202 (post-vaccination)
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 7 | 4 | 15 | 22 | 10 | 5
percentage of participants
  Day 91: number analyzed (Participants) | 7 | 7 | 4 | 0 | 0 | 0 | 0
  Day 91 | 71.4 [29.0 to 96.3] | 71.4 [29.0 to 96.3] | 25.0 [0.6 to 80.6] |  |  |  |
  Day 112: number analyzed (Participants) | 0 | 0 | 0 | 15 | 22 | 10 | 5
  Day 112 |  |  |  | 93.3 [68.1 to 99.8] | 90.9 [70.8 to 98.9] | 100 [69.2 to 100] | 40.0 [5.3 to 85.3]
  Day 181: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Day 181 | 100 [2.5 to 100] | 100 [2.5 to 100] |  |  |  |  |
  Day 202: number analyzed (Participants) | 0 | 0 | 0 | 1 | 12 | 0 | 0
  Day 202 |  |  |  | 100 [2.5 to 100] | 91.7 [61.5 to 99.8] |  |

23. Secondary Outcome: Number of Participants With Virologically-confirmed Coronavirus Disease (COVID-19)-Like Illness
Description: Virologically-confirmed COVID-19-like illness was defined by specified clinical symptoms and signs and confirmed by positive result for SARS-CoV-2 by nucleic acid amplification test (NAAT) on a respiratory sample in association with a COVID-19-like illness.
Time Frame: Cohort 1: up to Day 366 (post-vaccination) and Cohort 2: up to Day 387 (post-vaccination)
Population: Data was not collected and analyzed for this OM (virologically confirmed COVID-19 like illness) due to discontinuation of the development of the messenger ribonucleic acid (mRNA) COVID-19 vaccine by Sponsor. Hence, no further corresponding testing was conducted, and the planned efficacy analysis was not performed.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Serologically-confirmed SARS-CoV-2 Infection
Description: Serologically-confirmed SARS-CoV-2 infection as defined by SARS-CoV-2 Nucleoprotein specific antibody detection immunoassay was reported in this outcome measure.
Time Frame: Cohort 1: up to Day 366 (post-vaccination) and Cohort 2: up to Day 387 (post-vaccination)
Population: Data was not collected and analyzed for this OM (serologically confirmed SARS-CoV-2 infection) due to discontinuation of the development of the mRNA COVID-19 vaccine by Sponsor. Hence, no further corresponding testing was conducted, and the planned efficacy analysis was not performed.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Correlates of Risk/Protection Based on Antibody Responses to SARS-CoV-2
Description: Correlate of risk / protection based on antibody responses to SARS-CoV-2 was evaluated using virus neutralization or ELISA, considering virologically-confirmed COVID-19-like illness and/or serologically-confirmed SARS-CoV-2 infection.
Time Frame: Cohort 1: up to Day 366 (post-vaccination) and Cohort 2: up to Day 387 (post-vaccination)
Population: Data was not collected and analyzed for this OM (Correlates of Risk / Protection Based on Antibody Responses to SARS-CoV-2) due to discontinuation of the development of the mRNA COVID-19 vaccine by Sponsor. Hence, no further corresponding testing was conducted, and the planned efficacy analysis was not performed.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Group 3: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: Group 5: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected within 21 days post-vaccination. Solicited reaction data were collected within 7 days post any vaccination. SAE data were collected from Day 1 up to 12 months post last vaccination (i.e., up to Day 366 for Cohort 1 groups and up to Day 387 for Cohort 2 groups)
Description: SafAS population. In AE section, SR, Fever was reported as Pyrexia. AEs were planned to be collected & analyzed for combined population in which the same dose-level groups in Sentinel & FEC were pooled for analysis. One participant of Sentinel Cohort (ultra-low dose) who was supposed to receive 2 doses received only 1 ultra-low dose and thus was counted into Cohort 1: ultra-low dose (N = 37; 1 from sentinel cohort and 36 from FEC cohort 1) based on actual injection scheme.
Arm/Group | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 1: SARS-CoV-2 Vaccine Low Dose | Cohort 1: Placebo | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose | Cohort 2: SARS-CoV-2 Vaccine Low Dose | Cohort 2: SARS-CoV-2 Vaccine Medium Dose | Cohort 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/34 | 0/18 | 0/36 | 0/36 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/34 | 1/18 | 0/36 | 0/36 | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 31/37 | 30/34 | 11/18 | 34/36 | 35/36 | 10/10 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose (N=37) | Cohort 1: SARS-CoV-2 Vaccine Low Dose (N=34) | Cohort 1: Placebo (N=18) | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose (N=36) | Cohort 2: SARS-CoV-2 Vaccine Low Dose (N=36) | Cohort 2: SARS-CoV-2 Vaccine Medium Dose (N=10) | Cohort 2: Placebo (N=9)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: SARS-CoV-2 Vaccine Ultra Low Dose (N=37) | Cohort 1: SARS-CoV-2 Vaccine Low Dose (N=34) | Cohort 1: Placebo (N=18) | Cohort 2: SARS-CoV-2 Vaccine Ultra Low Dose (N=36) | Cohort 2: SARS-CoV-2 Vaccine Low Dose (N=36) | Cohort 2: SARS-CoV-2 Vaccine Medium Dose (N=10) | Cohort 2: Placebo (N=9)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 14 (14) | 17 (17) | 4 (4) | 20 (32) | 29 (48) | 9 (15) | 1 (1)
Injection Site Erythema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 5 (9) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 28 (28) | 28 (28) | 5 (5) | 33 (57) | 33 (64) | 10 (20) | 2 (3)
Injection Site Swelling (General disorders) | 1 (1) | 2 (2) | 0 (0) | 6 (7) | 4 (5) | 2 (3) | 0 (0)
Malaise (General disorders) | 21 (21) | 21 (21) | 5 (5) | 28 (47) | 31 (56) | 10 (18) | 2 (4)
Pyrexia (General disorders) | 5 (5) | 8 (8) | 1 (1) | 10 (14) | 16 (23) | 10 (18) | 0 (0) — Fever/Pyrexia events which occurred 7 days post-vaccination was considered as an unsolicited AE.
Covid-19 (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sars-Cov-2 Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (13) | 2 (2) | 20 (28) | 23 (37) | 10 (12) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (20) | 23 (23) | 4 (4) | 28 (45) | 28 (49) | 8 (15) | 2 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 18 (18) | 7 (8) | 26 (44) | 31 (55) | 10 (16) | 5 (6) — Headache events which occurred 7 days post-vaccination was considered as an unsolicited AE.
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early termination of this study by the Sponsor prior to full enrollment, the corresponding testing was not conducted, and few planned efficacy outcome measures data were not collected and analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04798027/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04798027/SAP_001.pdf